CLINICAL TRIAL: NCT03108235
Title: HOMe-based HEart Failure Self-Management Programme Study (The HOM-HEMP Study): A Randomized Controlled Trial
Brief Title: HOMe-based HEart Failure Self-Management Programme Study (The HOM-HEMP Study)
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: National University of Singapore (Other)
Collaborators: National University Hospital, Singapore (Other)
Responsible Party: Principal Investigator, Wang Wenru, Assistant Professor, National University of Singapore
Allocation: Randomized | Model: Parallel | Masking: Single | Purpose: Other
Other Study IDs: HSRGWS16Jul007
Record Dates: First submitted 2017-03-30; First posted 2017-04-11 (Actual); Last update posted 2021-03-15 (Actual); Status verified 2021-03

CONDITIONS: Heart Failure
Keywords: HF self-care; Multicomponent intervention; mHealth; Psychosocial education intervention
MeSH Terms: conditions — Heart Failure | interventions — Standard of Care

STUDY DESIGN:
Who Masked: Participant
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (3):
- Intervention group A (Experimental): a 6-week nurse-led, home-based self-management psychosocial education programme (HOM-HEMP)
  Interventions: Behavioral: HOM-HEMP
- Intervention group B (Experimental): HOM-HEMP with the smartphone app.
  Interventions: Behavioral: HOM-HEMP with smartphone app
- control group (Active Comparator): Participants will receive the standard care provided by the hospital. It consists of all nursing, medical, and follow-up services as needed.
  Interventions: Behavioral: Standard Care

INTERVENTIONS:
Behavioral: HOM-HEMP — a 6-week nurse-led, home-based self-management psychosocial education programme comprising of a specifically developed HF education and self-management toolkit, three biweekly home visits by the research nurse.
  Arms: Intervention group A
Behavioral: HOM-HEMP with smartphone app — a 6-week nurse-led, home-based self-management psychosocial education programme comprising of a specifically developed HF education and self-management toolkit, three biweekly home visits by the research nurse. In addition, participants will receive a smartphone app.
  The smartphone will be used to monitor their health data (such as weight, and blood pressure). The data will be synchronized to a web-connected portal on a remote server. The research nurse would be able to access your data through the web-connected portal and provide consultation through scheduled tele or video conference.
  Arms: Intervention group B
Behavioral: Standard Care — standard care provided by the hospital. It consists of all nursing, medical, and follow-up services as needed.
  Arms: control group

SUMMARY:
Aim: To develop a nurse-led, home-based self-management psychosocial education programme, entitled HOMe-based HEart Failure Self-Management Programme (HOM-HEMP), and evaluate its effects on improving heart failure self-care, cardiac self-efficacy, health-related quality of life (HRQoL), psychological well-being, perceived social support, and clinical outcomes among patients with heart failure in Singapore.

Background: The number of elderly people is expected to increase in the coming decades, and so too the prevalence of with chronic heart failure (HF) is expected to increase. Since HF is a chronic condition, there is a need to develop programmes that will improve the quality of life of older patients who have to manage this condition for years to come.

Design: A stratified, three-arm randomised controlled trial (RCT) will be adopted.

Methodology:

The HOM-HEMP is designed a six-week home-based psychosocial education programme comprising of a specifically developed HF education and self-management toolkit and three biweekly home visits by the research nurse. In addition, participants in experimental group B will receive a supplementary smartphone app.

A consecutive sample of 213 patients with HF will be recruited from the cardiac ward of a tertiary public hospital in Singapore. They will be randomly assigned to the control group, or experimental group A (HOM-HEMP without App) or the experimental group B (HOM-HEMP with App). A research nurse will be delivering the HOM-HEMP intervention to the participants in the experimental groups, while another research assistant who is blinded to participants' group assignment will be responsible for data collection.

Data will be collected at baseline, at 6 weeks from baseline (i.e. immediate after the intervention), and at 3 and 6 months from the baseline. At the end of the programme, a process evaluation will be conducted to assess the acceptability, strengths and weaknesses of the HOM-HEMP based on the participants' perspectives.

Discussion: It is expected the proposed RCT will make a contribution to knowledge development of the effectiveness of the HOM-HEMP and the active ingredients of the programme.

DETAILED DESCRIPTION:
Specific Aims

The primary aims of this study are:

1. To develop a nurse-led, home-based self-management psychosocial education programme, entitled HOMe-based HEart Failure Self-Management Programme (HOM-HEMP)
2. To examine its effectiveness on improving HF self-care, cardiac self-efficacy, anxiety and depression levels, health-related quality of life (HRQoL), perceived social support, and clinical outcomes among patients with HF in Singapore.

Study Hypotheses

Study participants will be randomised into one of the three groups: a Control Group (receiving usual care), an Experimental Group A (receiving HOM-HEMP without a supplementary smartphone App), and an Experimental Group B (receiving HOM-HEMP with a supplementary smartphone App).

It is hypothesised that participants in the Experimental Group A or B as compared with participants in the Control Group will have significantly:

1. Better HF self-care
2. Better cardiac self-efficacy.
3. Lower levels of anxiety and depression
4. Better HRQoL
5. Better perceived social support.
6. Better clinical outcomes, including improved NYHA functional class, and less unplanned health service utilization (i.e. unplanned medical consultation, emergency department visit due to heart disease, and hospital readmissions due to heart disease).

Approach adopted in the development of HOMe-based HEart Failure Self-Management Programme (HOM-HEMP).

The HOM-HEMP, is designed as a six-week home-based psychosocial education programme comprising of a specifically developed HF education and self-management toolkit and three biweekly home visits by the research nurse. The duration of the programme is determined based on the literature, in which the psychosocial interventions for patients with HF varied from two to 16 weeks across studies, with the average length being six weeks. In addition, participants in Experimental Group B will receive a supplementary smartphone app.

HOM-HEMP Education and Self-Management Toolkit Development

The toolkit will be developed for the participants to use whenever they encounter problems related to their condition at home. Participants can always read the education manual in the toolkit by themselves or with their family members/caregivers repeatedly to reinforce the learning of key information. The toolkit is therefore an important element of the whole programme.

The development of the content of the toolkit will follow patient-centred principle, which will be driven by patients' needs. The results of our recent study exploring the needs and living experiences of patients with HF in Singapore will be used to guide the research team to develop the toolkit. This is an important part of the development of the toolkit because it is crucial to ensure that the information presented is updated and relevant for local patients. This will help patients to make the necessary changes (e.g. healthier local food options instead of their current unhealthy choices) in their lifestyle, which is a key part of the recovery process. Another key emphasis of the development of the HF education manual is the psychosocial-related content which includes relaxation techniques, stress management, family and social support, and symptoms monitoring (e.g. shortness of breath, angina).The content of the HOM-HEMP education manual will include: (1) HF facts (e.g. definition, risk factors, signs and symptoms), and self-care principles, (2) stress and anxiety management (e.g. stress coping strategies, relaxation techniques), (3) medication management (e.g. effects and side-effects of medication), (4) physical exercises, (5) dietary and fluid management including practice tips, (6) smoking cessation (for smokers), and (7) family and social support (for family members and caregivers).

A panel of experts will be invited to validate the content of the toolkit to ensure it is relevant and helpful. The panel will include cardiologist, cardiac advanced practice nurse (APN), cardiac case manager, and one researcher who have experience in developing and running psychosocial education programmes. Special attention on the readability of the manual for older people will be considered when we design the manual, e.g. large-type print, short sentences, avoidance of medical terminology and jargon. Two lay HF patients will be also invited to review the drafted content. It is assuming that the educational level of most potential users would be at the lower end of reading skill required the easy use of written material.

HOM-HEMP Smartphone App Development

A smartphone app will be developed by a team of software engineers from School of Computing, National University of Singapore. The content and scope of the app will be mainly guided based on the content of the toolkit. The proposed functions included in the app are: (1) visual material including video clips of educational talks given by heart experts (e.g. triggering factors of CHF, signs and symptoms of CHF), relaxation techniques (e.g. deep breathing, meditation, muscle relaxation), stress management techniques (e.g. stress alleviating exercise) and recommended physical exercises (e.g. walking exercise, exercise logs) and Dietary matters (e.g. practical tips of selecting food, healthy recipes to try); (2) fluid calculator, (3) individualized scheduled reminders for doing exercise and relaxation, taking medication, medical appointment; salt/fluid targets; (4) weight/vitals logs (e.g. weight monitor, blood pressure and heart rate monitor with the use of Bluetooth-enabled devices such as Polar H7 or Wahoo Tickr) and (5) chat room with the research nurse.

The app will be designed as "elderly friendly" with features like large font size, using videos and pictures, and sound/voice reminders. There will be a monitoring function when participants log in the system. After the development of the app, it will be uploaded to mobile app stores, and users can download it from Googleplay (for Android users) or Apple app store (for IOS user) Technical issues such as compatibility, ease of use, potential causes of crashes will be tested. Once the test is completed, a field test will be conducted with 5 participants and/or their caregivers. They will be required to provide their overall evaluation of the app, and their feedback regarding the utilization of the app will guide the study team to further revise the app.

Study Design, Setting and Participants

A stratified randomised controlled, three-arm, pretest and repeated posttest design will be used in this project with both quantitative and qualitative measures. The study will be conducted at the cardiac ward of one of the largest acute public hospitals in Singapore. After the baseline measurements, the participants will be randomly assigned to one of the three groups using stratified randomization. These three groups are: the Control Group, in which participants will receive usual care; the Experimental Group A, in which participants will receive usual care and the HOM-HEMP intervention but without the supplementary smartphone app; the Experimental Group B, in which participants will receive the usual care, the HOM-HEMP intervention and the supplementary smartphone app.

One research nurse (RN) will be trained to conduct the intervention, and another research assistant (RA) will conduct the data collection. The RN will be responsible for delivering the HOM-HEMP to the participants (i.e. intervention), while the RA will be responsible for data collection. The RA will be blinded to participants' group assignment to prevent subjective bias stemming from the knowledge of grouping.

Four measurements will be conducted at the baseline prior to the intervention (T0), at 6 weeks from baseline, i.e. immediate after the intervention (T1), at 3 months from the baseline (T2), and at 6 months from the baseline (T3).

Outcome measures

Outcome measures include: Self-Care of Heart Failure Index (SCHFI), Cardiac Self-efficacy Scale (CSS), Hospital Anxiety and Depression Scale (HADS), Minnesota Living with Heart Failure Questionnaire (MLCHFQ), Short Form of the Social Support Questionnaire (SSQ6), NYHA Functional Classification, and unplanned Health service use.

Data will be collected at 6 weeks (immediate after the intervention), 3 months and 6 months from baseline.

Data analysis

The IBM SPSS 24.0 will be used for data analysis. Baseline categorical demographic characteristics across the 3 groups will be examined using Chi-squared or Fisher's Exact test; quantitative variables using ANOVA if normality and homogeneity assumptions satisfied otherwise Kruskal Wallis test will be used. General Linear Mixed Model (GLM) will be used to compare the study outcomes between 2 intervention groups against the Control group using Dunnett test at each individual time point. To correct for type 1 error on the multiple comparisons for each time point, statistical significance is set at p < 0.01. For the differences in the unplanned health service use between the experimental two groups against the control group, logistic regression will be performed adjusting for relevant covariates. A repeated measurement analysis will be performed to analyse the trend of groups' numerical outcomes over time setting significance level at p<0.05 and at two-tailed test.

For all qualitative data obtained from the face-to-face interviews, all audio taped interviews will be transcribed verbatim. Latent content analysis, which involves an interpretative reading of the symbolism underlying the surface structure in the text, will be used for the qualitative data-set. There are three basic steps involved in content analysis namely, developing meaningful units, developing the set of categories, and developing the rational and illustration to guide the coding of data into categories. This principle will guide the researcher to analyze the qualitative data gained from the interviews.

ELIGIBILITY:
Inclusion Criteria:

1. Clinically diagnosed with HF
2. 21 years or older, which is the legal age to give consent in Singapore
3. able to comprehend Chinese or English;
4. possess and able to use smart mobile phone (e.g. Samsung Galaxy, iPhone) in their daily lives, and
5. able to be followed up at home after hospital discharge.

Exclusion Criteria:

1. have unstable angina, resting tachycardia (>120 beats/minute), or severe arterial hypertension;
2. have a terminal illness other than HF, e.g. end-stage renal failure, cancer, severe pulmonary disease;
3. have psychiatric or cognitive impairment that will affect patient's understanding of the study intervention and/or nature of the study
4. are bed-bound or wheelchair-bound that will affect patient's ability to perform self-care
5. No internet access at home

Min Age: 21 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 213 (Actual)
Dates: Start 2018-06-01 (Actual); Primary Completion 2020-02-28 (Actual); Study Completion 2020-02-28 (Actual)

PRIMARY OUTCOMES:
HF self care | Data will be collected prior to the commencement of the programme (baseline), at 6 weeks, 3 months and again at 6 months from baseline
  As measured by the Self-Care Heart Failure Index (SCHFI)

SECONDARY OUTCOMES:
Cardiac Self-Efficacy | Data will be collected prior to the commencement of the programme (baseline), at 6 weeks, 3 months and again at 6 months from baseline
  Self-efficacy will be assessed by the Cardiac Self-efficacy Scale (CSS).
Anxiety and depression levels | Data will be collected prior to the commencement of the programme (baseline), at 6 weeks, 3 months and again at 6 months from baseline
  As measured by the Hospital Anxiety and Depression Scale (HADS).
Health-related quality of life (HRQoL) | Data will be collected prior to the commencement of the programme (baseline), at 6 weeks, 3 months and again at 6 months from baseline
  The HRQoL will be assessed by the Minnesota Living with Heart Failure Questionnaire (MLHFQ).
Perceived social support | Data will be collected prior to the commencement of the programme (baseline), at 6 weeks, 3 months and again at 6 months from baseline
  The social support will be measured using Short Form of the Social Support Questionnaire (SSQ6).

OTHER OUTCOMES:
NYHA Functional Classification | Data will be collected prior to the commencement of the programme (baseline), at 6 weeks, 3 months and again at 6 months from baseline
  The New York Heart Association (NYHA) functional classification.
Unplanned Health Service Use | Data will be collected at 6 weeks, 3 months and 6 months from baseline after the study intervention
  Unplanned health service use, including heart-related hospital readmission, visits to the emergency department, and medical consultation, will be assessed. The participants will be asked to indicate the number of times they have made unplanned use of health.
Semi-structured Interview-Process Evaluation | 6 months from baseline after participants complete the study
  The purpose of the semi-structured interview is to further assess the acceptability, strengths and weaknesses of the HOM-HEMP intervention based on the participants' perspectives.

CONTACTS AND LOCATIONS:
Overall Officials: Wenru Wang, PhD, Principal Investigator — National University of Singapore
Locations (1):
- National University of Singapore, Singapore, Singapore

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Derived] Jiang Y, Koh KWL, Ramachandran HJ, Nguyen HD, Lim S, Tay YK, Shorey S, Wang W. The effectiveness of a nurse-led home-based heart failure self-management programme (the HOM-HEMP) for patients with chronic heart failure: A three-arm stratified randomized controlled trial. Int J Nurs Stud. 2021 Oct;122:104026. doi: 10.1016/j.ijnurstu.2021.104026. Epub 2021 Jun 30. PMID 34271265